CLINICAL TRIAL: NCT04752020
Title: Prospective Assessment of Whether Adjuvant Netarsurdil Use Improves Post-Operative Outcomes in Patients Undergoing Descemetorhexis Without Endothelial Keratoplasty
Brief Title: Netarsudil Use After Descemtorhexis Without Endothelial Keratoplasty
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Emma C. Davies, MD, Principal investigator, Massachusetts Eye and Ear Infirmary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020P002755
Record Dates: First submitted 2021-02-02; First posted 2021-02-12 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Fuchs' Endothelial Dystrophy
Keywords: Descemetorhexis without endothelial keratoplasty
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Netarsudil use (Experimental): Patients will receive Netarsudil eye drops to use 1 drop nightly in the operative eye after DWEK surgery until corneal clearance
  Interventions: Drug: Netarsudil Ophthalmic

INTERVENTIONS:
Drug: Netarsudil Ophthalmic — Use of netarsudil after Descemetorhexis without endothelial keratoplasty

SUMMARY:
This will be a prospective assessment of whether adjuvant Netarsudil use in patients undergoing Descemetorhexis without endothelial keratoplasty improves time to corneal clearance and post-operative central endothelial cell counts. The anticipated enrollment is 25 patients.

DETAILED DESCRIPTION:
Subjects meeting inclusion criteria will be identified by Massachusetts Eye and Ear cornea surgeons during their pre-operative assessment and invited to participate in the study. Written informed consent will be obtained from the patient. The patients will then be added to a shared Epic patient list with a shared to-do column (outside of the patient record) indicating their subject ID and date of recruitment. All subjects will be asked to provide their best contact phone number which will be updated in the chart.

Upon obtaining informed consent, subjects will receive a bottle of Netarsudil from the Massachusetts Eye and Ear research pharmacy with post-operative instructions to use the drop once a day at bedtime starting on post-operative day 1 . Each patient will then receive regular, scheduled post-operative monitoring with a post-operative day 1 visit, post-operative week 1 visit, post-operative month 1 visit, and then every 2 month follow up for twelve months. Clinical examination, including best corrected visual acuity and intraocular pressure, will be recorded during every visit. Corneal topography and specular microscopy will be performed during the pre-operative assessment and during each bi-monthly visit in order to monitor for post-operative outcomes.

A retrospective chart review will be performed prior to new patient enrollment for patients who had previously had DWEK and did not receive a rho-kinase inhibitor. These patients will be included for pre-operative and post-operative vision, pachymetry, corneal topography results, and specular microscopy results with minimization of data acquisition as no informed consent can be obtained from these patients.

ELIGIBILITY:
Inclusion Criteria:

* Fuchs corneal dystrophy

Exclusion Criteria:

* Women of childbearing potential
* Other corneal eye diseases
* Non-compliance with netarsudil
* Intolerance of netarsudil

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-03-28 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Change in central corneal pachymetry over time | Measured at post-operative month one visit and then every 2 months for 1 year
  Corneal thickness on clinical examination and corneal topography
Change in endothelial cell count over time | Measured at post-operative month one visit and then every 2 months for 1 year
  Central endothelial cell count by specular microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Emma Davies, MD, Principal Investigator — Massachusetts Eye and Ear Infirmary; Sila E Bal, MD, MPH, Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bal S, Pineda R, Davies E. Prospective Assessment of Adjuvant Netarsudil Use in Patients Undergoing Descemet Stripping Only. Cornea. 2025 Mar 1;44(3):286-290. doi: 10.1097/ICO.0000000000003578. Epub 2024 May 23. PMID 38780446